CLINICAL TRIAL: NCT01007760
Title: Dose-dependent Biological Mechanisms of Second-hand Smoke on Endothelial Function and Oxidative Stress
Brief Title: Dose-dependent Effects of Second-hand Smoke on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Peter Ganz, M.D., UCSF
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TRDRP-18FT-0049
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Disease
Keywords: Tobacco smoke; Oxidative stress; Endothelial Function; Atherosclerosis; Arterial Stiffness; Microvascular Function
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis | interventions — Tobacco Smoke Pollution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Room air (Placebo Comparator)
  Interventions: Other: Respirable suspended particles (RSP) PM 2.5 dose of second-hand smoke
- Low dose exposure second-hand smoke (Active Comparator)
  Interventions: Other: Respirable suspended particles (RSP) PM 2.5 dose of second-hand smoke
- High dose exposure second-hand smoke (Active Comparator)
  Interventions: Other: Respirable suspended particles (RSP) PM 2.5 dose of second-hand smoke

INTERVENTIONS:
Other: Respirable suspended particles (RSP) PM 2.5 dose of second-hand smoke — acute one time exposure

SUMMARY:
The purpose of this study is to determine the vascular effects of brief second-hand smoke exposure on normal healthy individuals.

DETAILED DESCRIPTION:
Second-hand smoke remains a significant public health threat. Despite evidence to suggest that secondhand smoke contributes to adverse cardiovascular outcomes, little is known about the dose-dependent vascular effects of brief secondhand smoke exposure at low doses commonly encountered in the community. This study will investigate the acute vascular effects and dose-dependent biological mechanisms of secondhand smoke on endothelial function and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking adults

Exclusion Criteria:

* Reported Active Smoking
* History of diabetes, hypertension, chronic respiratory disease, coronary artery disease, prior myocardial infarction or heart failure
* Pregnancy or breastfeeding
* Current use of prescription drugs within 14 days of trial
* Reported significant passive smoke exposure or elevated cotinine levels

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Flow-mediated dilation (FMD) | Same day - before/after exposure

SECONDARY OUTCOMES:
Plasma measurement of asymmetric dimethylarginine (ADMA) and Nitrotyrosine levels | Same day - before/after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ganz, MD, Principal Investigator — UCSF San Francisco General Hospital
Locations (1):
- UCSF San Francisco General Hospital, San Francisco, California, United States